CLINICAL TRIAL: NCT03813836
Title: A Phase II Trial to Assess the Efficacy and Safety Profile of Pembrolizumab in Patients With Performance Status 2 With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Phase II Trial of Pembrolizumab in Recurrent or Metastatic HNSCC
Acronym: POPPY
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/17/0396
Record Dates: First submitted 2019-01-15; First posted 2019-01-23 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Head and Neck Squamous Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma
Keywords: Head and Neck Cancer; Metastatic Head and Neck Squamous Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma; Pembrolizumab
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pembrolizumab + best supportive care (Experimental): Best supportive care and pembrolizumab 200mg every 3 weeks for a maximum duration of 24 months
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Patients will receive best supportive care + pembrolizumab 200mg every 3 weeks for a maximum duration of 24 months
  Other Names: Keytruda

SUMMARY:
A single-arm phase II trial to assess the efficacy and safety profile of pembrolizumab in patients with performance status of 2 with recurrent or metastatic squamous cell carcinoma of the head and neck. Patients will receive best supportive care + pembrolizumab 200mg every 3 weeks for a maximum duration of 24 months

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed locally advanced, recurrent or metastatic squamous cell carcinoma of the head and neck that is considered incurable by local therapies
2. Measurable disease evaluated by RECIST criteria version 1.1
3. WHO performance status of 2
4. Life expectancy >12 weeks
5. Aged ≥18 years of age
6. Adequate bone marrow function
7. Adequate renal function
8. Adequate liver function
9. Willing to use highly effective contraception for the duration of trial treatment and for 120 days after completion of treatment
10. Able to give informed consent, indicating that the patient has been informed of and understands the experimental nature of the study, possible risks and benefits, trial procedures, and alternative options
11. Willing and able to comply with the protocol for the duration of the study, including the treatment plan, investigations required and follow up visits

Exclusion Criteria:

1. Patients with undifferentiated nasopharyngeal or sino-nasal cancers
2. Disease suitable for treatment with curative intent
3. Prior therapy with an anti-PD-1, anti-PD-L1 or anti-PD-L2 agent
4. Any investigational agents within 4 weeks prior to registration
5. Anti-cancer monoclonal antibody therapy within 4 weeks prior to registration
6. Chemotherapy, targeted small molecule therapy, or radiotherapy within 2 weeks prior to registration
7. Patients with concurrent or previous malignancy that could compromise assessment of the primary or secondary endpoints of the trial
8. Women who are pregnant or breast feeding
9. Grade 3 or 4 peripheral neuropathy
10. Any serious and/or unstable pre-existing medical, psychiatric or other condition that, in the treating clinician's judgment, could interfere with patient safety or obtaining informed consent
11. Active central nervous system (CNS) metastases and/or carcinomatous meningitis
12. Active hepatitis B or C infection
13. Immunocompromised patients (e.g. known HIV positive status)
14. Prior organ transplantation including allogenic stem-cell transplantation
15. History of (non-infectious) pneumonitis/interstitial lung disease that required steroids, or current pneumonitis/interstitial lung disease
16. Active infection requiring systemic therapy
17. Received a live vaccine within 30 days prior to registration
18. Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
19. Active autoimmune disease that might deteriorate when receiving an immune-stimulatory agent.
20. Current use of immunosuppressive medication (exceptions apply) Refer to section 7.2 for full list of eligibility criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Disease control rate at 24 weeks assessed using iRECIST | 24 weeks after registration
  Disease control rate (proportion of patients with CR, PR or SD) assessed using iRECIST

SECONDARY OUTCOMES:
Disease control rate assessed using iRECIST | 12 months after registration
  Disease control rate (proportion of patients with CR, PR or SD) assessed using iRECIST
Best Response Rate- measured using the change from baseline tumour size. Assessed using iRECIST. | 6 months after registration
  Best Response Rate, defined as proportion of patients who have a CR or PR as their best response, measured using the change from baseline tumour size, assessed using iRECIST
Clinical Benefit Rate -defined as patient's best response rate lasting at least 18 weeks | From start of treatment to 30 months post start of treatment
  Clinical Benefit Rate, defined as proportion patients who have achieved CR, PR or SD as their best response lasting at least 18 weeks
Duration of Response- defined as the time from first documented evidence of CR or PR until disease progression or death. | From start of treatment to 30 months post start of treatment
  Duration of Response, defined as the time from first documented evidence of CR or PR until disease progression or death
Time to Progression -defined as time from registration to the first documented disease progression | From registration to 30 months post start of treatment
  Time to Progression, defined as time from registration to the first documented disease progression
Progression Free Survival defined as the time from registration to the first documented disease progression or death due to any cause, whichever occurs first. | From registration to 30 months post start of treatment
  Progression Free Survival, defined as the time from registration to the first documented disease progression or death due to any cause, whichever occurs first.
Overall Survival- defined as the time from registration to death due to any cause. | From registration to 30 months post start of treatment
  Overall Survival, defined as the time from registration to death due to any cause.
Frequency and severity of adverse events- throughout the patient's treatment and until 6 months after completion of trial treatment. | From date of registration until 6 months after completion of trial treatment
  Frequency and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Martin Forster, FRCP PhD, Principal Investigator — University College, London
Locations (12):
- United Kingdom (12):
  - Aberdeen Royal Infirmary (NHS Grampian), Aberdeen
  - Bristol Haematology and Oncology Centre (University Hospital Bristol NHS Foundation Trust), Bristol
  - Western General Hospital (NHS Lothian), Edinburgh
  - East Suffolk and North Essex NHS Foundation Trust, Ipswich
  - Guy's and St Thomas' NHS Foundation Trust, London
  - University College London Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral
  - East and North Hertfordshire NHS Trust, Northwood
  - Queens Hospital (Barking, Havering and Redbridge University Hospitals NHS Trust), Romford
  - Musgrove Park Hospital (Somerset NHS Foundation Trust), Taunton
  - Royal Cornwall Hospital Trust, Truro